CLINICAL TRIAL: NCT03052777
Title: Improving Quality of Life in Hematologic Cancer Survivors by Closing the Exercise Intention-Behavior Gap: a Phase II Randomized Controlled Trial of a Theory-based, Telephone-delivered Exercise Counselling Intervention
Brief Title: Using Telephone Counselling to Improve Exercise Participation in Hematologic Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Kerry Courneya, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-16-0775
Record Dates: First submitted 2017-01-31; First posted 2017-02-14 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Leukemia; Lymphoma; Lymphoma, Non-Hodgkin; Behavior, Health
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Non-Hodgkin; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Counselling (Experimental): Participants will be asked to increase their exercise by at least 60 minutes per week and will receive a copy of Canada's Physical Activity Guideline plus 12 weekly telephone counseling sessions aimed at helping survivors follow-through on their exercise intention.
  Interventions: Behavioral: Telephone counselling
- Control (No Intervention): Participants will be asked to increase their exercise by at least 60 minutes per week and will be self-directed, only receiving a copy of Canada's Physical Activity Guideline as standard of care.

INTERVENTIONS:
Behavioral: Telephone counselling — The intervention is a 12 week telephone counselling exercise program where participants will receive weekly telephone counselling that targets key theoretical behavior change constructs. Participants will also receive a copy of Canada's Physical Activity Guideline.
  Arms: Telephone Counselling

SUMMARY:
This study evaluates the impact of a 12-week theory-based exercise telephone counselling program (versus a self-directed exercise group) on closing the exercise intention-behavior gap in a sample of hematologic cancer survivors.

DETAILED DESCRIPTION:
Problem: Regular exercise participation improves quality of life and physical function for cancer survivors. Unfortunately, the most effective way of promoting exercise to cancer survivors has yet to be determined, and as a result, many survivors are inactive. Theory-based efforts have typically focused on promoting intentions to exercise, though we are now discovering that only about half of those who intend to exercise actually follow through on their intentions. This is known as the exercise intention-behavior gap. It also appears that survivors are more likely to follow-through on their intention to exercise when they report employing key behavioral and motivational strategies (i.e., creating detailed exercise plans, feeling capable and obligated to exercise, perceiving it to be beneficial and fun, and avoiding the temptation to participate in alternative activities) which may be promoted via telephone counselling.

Objective: To determine whether a theory-based telephone counselling intervention focused on closing the exercise intention-behavior gap is feasible and can improve exercise levels, motivation, quality of life, and fatigue in hematologic cancer survivors.

Methods: A two-armed randomized controlled trial will compare the efficacy of telephone counselling versus a control condition (self-directed with Canada's Physical Activity Guide). All participants will be asked to increase their exercise by at least 60 minutes per week. Hematologic cancer survivors who previously participated in an exercise survey study and indicated interest in participating in future exercise related research (N=407) will be contacted to participate in the current trial. Eligible participants will be randomized in a 1:1 ratio to either the telephone counseling group or a self-directed exercise group. Participants in the intervention arm will receive 12 weekly telephone counseling sessions aimed at helping survivors follow-through on their exercise intention. A sample of approximately N=66 hematologic cancer survivors will be recruited for this 12-week trial. Data will be collected via online surveys assessing changes in exercise levels, motivation, quality of life, and fatigue. Feasibility will be determined by eligibility percentage, recruitment percentage, adherence rate, assessment completion rate, adverse events, and ratings of program acceptability.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study will be survivors who have had a histologically confirmed hematologic cancer, and who are between 18-80 years of age, living in Alberta, can speak and comprehend English, and willing to participate in a 12-week exercise telephone counseling intervention.

Exclusion Criteria:

* Survivors reporting greater or equal to 150 minutes of moderate-to-vigorous exercise will be excluded because they will already be meeting the public health guidelines for exercise. Survivors planning to be away for more than 2 weeks during the intervention, or with major exercise contraindications will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Exercise Levels | Baseline and within 7 days of completing the 12-week intervention
  Exercise levels assessed using the Godin Leisure-Time Exercise Questionnaire

SECONDARY OUTCOMES:
Change from baseline in Exercise Motivation | Baseline and within 7 days of completing the 12-week intervention
  Exercise motivation assessed via validated questionnaires that align with the Multi-Process Action Control Framework
Change from baseline in Quality of life | Baseline and within 7 days of completing the 12-week intervention
  Quality of life assessed using the Short Form-36 (SF-36) questionnaire
Change from baseline in Fatigue | Baseline and within 7 days of completing the 12-week intervention
  Fatigue assessed using the Functional Assessment of Cancer Therapy: Fatigue (FACT-F) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vallerand JR, Rhodes RE, Walker GJ, Courneya KS. Social Cognitive Effects and Mediators of a Pilot Telephone Counseling Intervention to Increase Aerobic Exercise in Hematologic Cancer Survivors. J Phys Act Health. 2019 Jan 1;16(1):43-51. doi: 10.1123/jpah.2018-0014. Epub 2018 Dec 2. PMID 30501541
- [Derived] Vallerand JR, Rhodes RE, Walker GJ, Courneya KS. Feasibility and preliminary efficacy of an exercise telephone counseling intervention for hematologic cancer survivors: a phase II randomized controlled trial. J Cancer Surviv. 2018 Jun;12(3):357-370. doi: 10.1007/s11764-018-0675-y. Epub 2018 Feb 6. PMID 29411314